CLINICAL TRIAL: NCT05571943
Title: A Multicenter, Open-label Study to Assess the Long-term Safety of Difamilast Ointment 1% in the Treatment of Children, Adolescents and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: A Open-label Study to Assess the Long-term Safety of Difamilast Ointment 1% in Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM36-302
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Difamilast Ointment 1% (Experimental): A thin layer of Difamilast applied to affected areas twice daily (morning and evening, approximately 12 hours apart)
  Interventions: Drug: Difamilast

INTERVENTIONS:
Drug: Difamilast — Difamilast Ointment 1%

SUMMARY:
This is a Phase 3, open-label study to evaluate the long-term safety of difamilast ointment 1% in subjects ≥2 years of age with mild to moderate AD. The study will also evaluate the long-term efficacy of difamilast ointment 1%, including durability of response.

ELIGIBILITY:
Important Inclusion Criteria:

1. Subjects who are male or female ≥2 years of age at Screening (Visit 1).
2. Subjects who have a diagnosis of AD based on the American Academy of Dermatology AD diagnostic criteria
3. Subjects who have had a diagnosis of AD for at least 3 months prior to Screening .
4. Subjects who have an IGA of mild or moderate AD Severity and treatable body surface area (BSA) ≥3%at Baseline if not previously enrolled in study MEDI-MM36-301 OR b. IGA ≤ 3, with no minimum BSA and completed through Week 4/EOT Visit 6 of the study MEDI-MM36-301.
5. Subject is willing and able to comply with all study-related procedures, including, but not limited to, application of the study drug, and visit requirements.

Important Exclusion Criteria:

1. Subjects who have an AD flare (defined as rapid intensification of AD) within 28 days prior to Screening or Baseline (except for those previously enrolled in Study MEDI-MM36-301) or history of consistent requirement for high-potency topical corticosteroids to manage AD signs and symptoms.
2. Subjects who have an active or acute skin infection (eg, herpes simplex, herpes zoster, or chicken pox), and/or clinically infected AD
3. Subjects with significant systemic or localized infection
4. Subjects with minimal/mild depression and suicidal ideation
5. Subjects using restricted medications, biologics and alternative therapies, or using investigational drug

   -

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and their relationship to study drug | 52 week study period
Proportion of subjects who discontinue due to an AE over the study period | 52-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Uma S Atmuri, MPharm MS, Study Director — Acrotech Biopharma Inc.
Locations (63):
- United States (63):
  - Qualmedica Research, LLC, Birmingham, Alabama
  - AllerVie Health, Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - NEA Baptist Clinic-Dermatology, Jonesboro, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Southern CA Dermatology Skin and Laser, Laguna Niguel, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Clarity Dermatology, LLC, Castle Rock, Colorado
  - IMMUNOe Research Centers, Centennial, Colorado
  - TrueBlue Clinical Research, Brandon, Florida
  - Annexus Dermatology & Aethestics, DeLand, Florida
  - Accel Research - Edgewater Clinical Research Unit, Edgewater, Florida
  - Skin Care Research, Hollywood, Florida
  - Kirsch Dermatology, Naples, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Pure Skin Dermatology & Aesthetics, Orlando, Florida
  - Nona Pediatrics, Orlando, Florida
  - Accel Research - Ormond Clinical Research Unit, Ormond Beach, Florida
  - Olympian Clinical Research, St. Petersburg, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - Arlington Dermatology, Rolling Meadows, Illinois
  - DS Research, Clarksville, Indiana
  - Qualmedica Research, LLC, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Options Research Group, LLC, West Lafayette, Indiana
  - Meridian Clinical Research, Overland Park, Kansas
  - Qualmedica Research, LLC, Bowling Green, Kentucky
  - DS Research, Louisville, Kentucky
  - Clinical Trials Management, LLC, Covington, Louisiana
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - DermAssociates, LLC, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Oakland Hills Dermatology, PC, Auburn Hills, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Cleaver Dermatology, Kirksville, Missouri
  - Vivida Dermatology, Las Vegas, Nevada
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Bexley Dermatology Research, Bexley, Ohio
  - Optima Research, Boardman, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Optimed Research, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Peak Research, LLC, Upper Saint Clair, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Anderson, South Carolina
  - Coastal Pediatric Research, Charleston, South Carolina
  - International Clinical Research - Tennessee, LLC, Murfreesboro, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Derm Research, Austin, Texas
  - J&S Studies, College Station, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Center for Clinical Studies, Ltd, LLP, Houston, Texas
  - Research Your Health, Plano, Texas
  - Houston Center for Clinical Research, Sugar Land, Texas
  - Center for Clinical Studies, Webster, Texas
  - Premier Clinical Research, LLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No